CLINICAL TRIAL: NCT01623011
Title: What is the Clinical and Cost Effectiveness of Arthroscopic Sub-acromial Decompression Surgery?
Brief Title: Can Shoulder Arthroscopy Work
Acronym: CSAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Arthritis Research UK (Other); University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSAW
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder; Sub-acromial; Rotator Cuff; Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Arthroscopy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arthroscopic Sub-acromial Decompression (Experimental): Arthroscopic sub-acromial decompression surgery.
  Interventions: Procedure: Arthroscopic Sub-acromial Decompression Surgery
- Shoulder Arthroscopy (Active Comparator): Shoulder arthroscopy only.
  Interventions: Procedure: Shoulder Arthroscopy
- Active Monitoring with Specialist Reassessment (Other): Active monitoring with specialist reassessment - non-operative control.
  Interventions: Other: Active Monitoring with Specialist Reassessment

INTERVENTIONS:
Procedure: Arthroscopic Sub-acromial Decompression Surgery — The procedure involves insertion of the arthroscope into the glenohumeral joint where the joint surface is inspected along with the intra-articular portion of the long head of biceps and the joint surface of the rotator cuff tendons. The arthroscope is then inserted into the sub-acromial bursa which lies outside the rotator cuff tendons and beneath the acromion process of the scapula. In the bursa the acromion and superior surface of the rotator cuff are assessed to ensure the coracoacromial ligament and the AC joint remains intact. The projecting under surface of the distal part of the acromion is resected.
  Other Names: ASAD
  Arms: Arthroscopic Sub-acromial Decompression
Procedure: Shoulder Arthroscopy — This is the surgical comparison group. The procedure is performed under general anaesthetic. Patients will undergo a routine investigational arthroscopy. The operation will be performed in exactly the same manner as Group ASAD. The exception is they will not undergo the decompression (bone spur removal). Tissues will be visualised and the joint will be washed out. The time spent in theatre will be similar to that for Group ASAD. These measures provide the AO group with the characteristics necessary to provide a reasonable comparison and account for the placebo effects of surgery.
  Other Names: Arthroscopy alone
  Arms: Shoulder Arthroscopy
Other: Active Monitoring with Specialist Reassessment — Patients will be advised that they will undergo active monitoring in the short term. They will attend a reassessment appointment 3 months after entering the study. Here, they will be asked to complete questionnaires related to their shoulder pain and undergo a clinical assessment for their shoulder. From an ethical standpoint it is emphasised that it is quite within normal practice to have a period of active monitoring.
  Other Names: Non-operative group; Control group
  Arms: Active Monitoring with Specialist Reassessment

SUMMARY:
Shoulder problems causing pain and decreased function are very common. Many of these problems are related to the rotator cuff tendons. Shoulder arthroscopy surgery (keyhole surgery) is a common treatment for this pain. This can involve an Arthroscopic Subacromial Decompression (ASAD) an operation used to remove bony spurs which may be the cause of the pain. This procedure is widely used despite limited evidence of any effectiveness. This is a randomised controlled trial that will compare ASAD against an investigational shoulder arthroscopy (without spur removal/decompression) to indicate whether spur removal is really necessary and in turn, assessing the effectiveness of the ASAD procedure. Both surgical interventions are routine and will mirror each other except for the spur removal element. Both treatments will be compared against a control (non operative management with specialist reassessment) group to indicate whether surgery in general is effective for patients with subacromial pain. Patients randomised to either of the surgical options will be blinded to the type of surgery they have. This is a multicentre trial taking place in 10 centres in England and Wales. Two satellite studies will also take place. One will involve a subset of patients undergoing MRI scans to examine the effects of their shoulder pain on their brain transmissions. The other will involve collecting tissue samples from patients undergoing surgery.

DETAILED DESCRIPTION:
The prevalence of shoulder complaints in the UK is estimated to be 14%, with 1-2% of adults consulting their general practitioner annually regarding new-onset shoulder pain. Rotator cuff pathology, including rotator cuff tears and sub-acromial pain, reportedly accounts for up to 70% of shoulder pain problems. Other common causes of shoulder pain include frozen shoulder, calcific tendonitis and osteoarthritis (OA).

Painful shoulders pose a substantial socioeconomic burden. Disability of the shoulder can impair ability to work or perform household tasks and can result in time off work. Shoulder problems account for 2.4% of all general practitioner consultations in the UK and 4.5 million visits to physicians annually in the USA. With the exception of fractures and traumatic rotator cuff tears, most shoulder pain problems are treated initially with conservative care. In some patients with persistent symptoms, surgery might be required. More than 300,000 surgical repairs for rotator cuff pathologies are performed annually in the USA, and the annual financial burden of shoulder pain management in the USA has been estimated to be US$3 billion.

Sub-acromial pain is the most frequent cause of shoulder problems in the general population. An anatomical etiology has been proposed, whereby mechanical contact occurs between the rotator cuff tendons and the overlying acromion and coracohumeral ligament. Sub-acromial pain and rotator cuff tears are associated with progressive change in the shape of the acromion, with 'spurs' forming at its antero-inferior margin. Evidence suggests spurs develop which narrow the sub-acromial space, thereby making physical contact more likely, particularly in certain positions of the arm (for example, painful arc), and resulting in inflammation. This is sometimes referred to as "impingement". However this term suggests a definitive mechanism of the pain and conflicting theories indicate such mechanisms are not definitive. For the purposes of this study we will continue to refer to this as "sub-acromial pain".

A high proportion of patients with sub-acromial pain will respond to conservative treatment. The most frequent indications for surgery are persistent and severe pain combined with functional restrictions that are resistant to conservative measures. Despite surgery being considered at this point, some reports show that surgery can be no more effective than physiotherapy in the relief of pain when used in patients at this stage. Surgical intervention can, however, achieve good results and its judicious use seems valid. The most common surgical intervention for sub-acromial pain is a sub-acromial decompression (SAD), which can be performed through an arthroscopic (ASAD) approach. An assessment of the cost of treatment of impingement also suggested that the addition of surgery, in comparison to exercise treatment alone, is not cost-effective.

Further research might identify whether the source of pain is the tendon, the acromion or the bursa, and hence help to rationalize surgical treatment.

One possible sequela of sub-acromial pain is a rotator cuff tear. The term 'rotator cuff tear' refers to structural failure and tissue disruption in at least one of the four muscles and tendons that form the rotator cuff. Any tear that involves rotator cuff disruption that does not extend all the way through the tendon is termed a partial-thickness tear (PTT). PTTs are more prevalent than full-thickness tears. Information is lacking regarding the risk of progression of PTTs to full-thickness tears although it is thought that lesions involving less than 50% of the thickness of the cuff are at risk of progression in the long term as shown by Cordasco et al. The management of PTTs is controversial and patients with PTTs have commonly been treated conservatively. If the symptoms fail to resolve with conservative treatment then ASAD might be beneficial. Favourable results have been reported following debridement of PTT in association with ASAD.

It is largely assumed that arthroscopic sub-acromial decompression (ASAD) has some therapeutic benefit. This is on the assumption that much of the pain and symptoms of sub-acromial pain is due to mechanical contact between the upper surface of the rotator cuff tendons and the under-surface of the acromion. This pain is also believed to be associated with inflammation of the intervening sub-acromial bursa.

ASAD has been performed for the treatment of sub-acromial pain and rotator cuff disease for the last 35 years. The number of ASADs performed by orthopaedic surgeons has increased significantly over time. A fact made remarkable by the absence of any compelling or concrete evidence in support of the procedure. Recent figures from the USA report a 254% increase (from 29.9 to 102.2 per 100 000 people per year) in use of the procedure in New York State between 1996 and 2006 with only a 74% increase in orthopaedic surgery overall and a 475% increase (from 3.3 to 19.0 per 100 000 people per year) in use of the procedure in Olmsted County, Minnesota in the 25 years leading up to 2005. Although both studies show a significant increase in use of the procedure, the New York State surgeons perform over five times as many decompressions as their colleagues in Rochester Minnesota. The introduction of less invasive arthroscopic techniques accounts for some of the overall increased rate of surgery but does not explain the geographical variation. Patient and disease characteristics have not changed over time and there is a growing concern that this procedure is being overused. Observational studies of ASAD show positive results in terms of pain reduction and functional outcome with high patient satisfaction rates. However, equally good outcomes have been noted in two studies following patients who had arthroscopic rotator cuff debridement or open rotator cuff repair in the absence of a sub-acromial decompression. Furthermore, comparative studies of ASAD versus non-operative treatment options, such as physiotherapy, have not shown any significant difference in outcome between the two treatment modalities.

There are a growing number of studies that have tried to assess the effectiveness of sub-acromial decompression against a control. Two studies randomised patients undergoing rotator cuff repair to groups including or excluding sub-acromial decompression in their operative treatment, neither demonstrated any difference in outcome between the groups. In an important recently reported randomised controlled trial, ASAD plus sub-acromial bursectomy was compared with bursectomy alone and reported no significant difference in clinical outcome between the two groups. This finding suggests that removing acromial spurs might not be necessary.

These studies support the theory that undergoing a surgical intervention for sub-acromial pain carries a significant placebo effect and that removal of the sub-acromial spur of bone may not be necessary.

Unfortunately no randomised trials have been performed on patients with sub-acromial pain to show that ASAD is more effective than simply inserting the arthroscope, as per investigative arthroscopy, or doing nothing at all (no treatment). The NHS Database of Uncertainties about the Effects of Treatment (DUETs) confirms the lack of evidence. They highlight the low level of evidence available and the high susceptibility of bias which exists in some of the publications on this topic. Therefore, we remain ignorant of the mode of action for any potential therapeutic effect. All three options are yet to be tested satisfactorily.

To unequivocally state that surgery treatment is effective, the surgical procedure must be compared against a sham or placebo treatment. A sham surgery must be a mock up or imitation of the procedure. It is virtually impossible to imitate an operation without actually performing the surgery. In terms of placebo, there have been previous placebo controlled trials in surgery, particularly in the lower limb, with some interesting results. It is known that the very process of undergoing surgery (without necessarily affecting the structures involved in the pathology) can generate a beneficial outcome. This has been shown in the knee where a placebo controlled trial of arthroscopic surgery for osteoarthritis of the knee. This found that, despite early benefit, one year results after arthroscopic lavage or debridement were no better than after an entirely placebo operative procedure.

Psychological mechanisms of treatments can have meaningful therapeutic effects. These may include expectations, memory, motivation, somatic focus, reward, anxiety reduction and meaning. Expectancy requires patients to have expectations of future responses to treatment. Arguably surgery, with all its attendant verbal and non-verbal clues, is a very powerful modulator of expectancy and could therefore have a profound placebo effect.

Responses may also be conditioned and mediated through physiological changes in hormones and immune response. Most research into the neurobiology of placebo has investigated analgesia. Shoulder arthroscopy and sub-acromial decompression is principally (if not entirely) focused on relief of pain and patients undergoing this relatively low risk day case surgical procedure may well be affected by some form of placebo effect. Analgesic responses to placebo often involve endogenous opioid mechanisms. Other neuro-transmitters and neuromodulators may also be involved.

To consider the effects of such placebo potential, the surgical procedure in question should have the key mechanical element(s) of the operation isolated and omitted. In this way the therapeutic mechanisms of the surgery can be evaluated and any perceived or non-specific effects of the surgery can be highlighted.

ELIGIBILITY:
Inclusion Criteria:

* Sub-acromial pain of at least 3 month (tendinopathy and partial tear only).
* Diagnosed by a Consultant of tendinopathic pain or partial thickness rotator cuff tear
* Has had an MRI or Ultrasound Scan to rule out alternative pathology
* Eligible for surgery.
* Completed a conservative management programme previously including:

  * physiotherapy that includes a remedial exercise regimen and
  * at least x1 cortisone injection but not more than 3 injections.

Exclusion Criteria:

* Full thickness tear of the rotator cuff tendons evident on MRI or Ultrasound imaging
* Undergone previous surgery on affected shoulder
* Have RA or other inflammatory disorder
* Symptomatic cervical spine pathology
* Previous septic arthritis
* History of radiotherapy on same side as affected shoulder
* Patients who have a strong preference for one treatment over another to an extent that they would not participate if allocated to their non- preferred group.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2012-09-14 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 6 months post randomisation
  Patient reported outcome measure of shoulder pain and function.

SECONDARY OUTCOMES:
Oxford Shoulder Score | 12 months post randomisation
  Patient reported outcome measure of shoulder pain and function
Constant Murley Shoulder Score | 6 and 12 months post randomisation
  Clinical assessment of the shoulder
Pain DeTECT | 6 and 12 months post randomisation
  Patient reported outcome related to neuropathic pain
Quantitative Sensory Testing | 6 and 12 months post randomisation
  Clinical assessment of pain and pain thresholds
Health Economics - EQ5D | 6 and 12 months post randomisation
  Patient reported expenditure and quality of life questions
Complications | 6 and 12 months post randomisation
  Patient reported complications post randomisation
Treatment Expectations and Satisfaction | 6 and 12 months post randomisation
  Patient reported questions on treatment expectations and satisfaction with treatment.
Hospital Anxiety and Depression Scale | 6 and 12 months post randomisation
  Patient reported questionnaire related to their feelings of anxiety and depression.
Patient Response Shift | 12 months post randomisation
  patient response shift on perceived disability will be assessed by comparing each patients pre-operative self-evaluation of their disability (baseline Oxford Shoulder Score) with a 12 month evaluation of their perceived pre-intervention state (the "thentest") according to the method of Razmjou et al (2010. This will give an indication of whether patients with sub-acromial pain underrate or overrate their pre-intervention disability according to their outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David J Beard, Professor, Study Chair — University of Oxford; Andrew J Carr, Professor, Study Chair — University of Oxford; Jonathan Rees, Principal Investigator — University of Oxford; Jonathan Cook, Principal Investigator — University of Aberdeen; Irene Tracey, Principal Investigator — University of Oxford; Steven Gwilym, Principal Investigator — University of Oxford; Cushla Cooper, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Department of Orthopaedics, Rheumatology & Musculoskeletal Sciences, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Beard DJ, Rees JL, Cook JA, Rombach I, Cooper C, Merritt N, Shirkey BA, Donovan JL, Gwilym S, Savulescu J, Moser J, Gray A, Jepson M, Tracey I, Judge A, Wartolowska K, Carr AJ; CSAW Study Group. Arthroscopic subacromial decompression for subacromial shoulder pain (CSAW): a multicentre, pragmatic, parallel group, placebo-controlled, three-group, randomised surgical trial. Lancet. 2018 Jan 27;391(10118):329-338. doi: 10.1016/S0140-6736(17)32457-1. Epub 2017 Nov 20. PMID 29169668
- [Derived] Savulescu J, Wartolowska K, Carr A. Randomised placebo-controlled trials of surgery: ethical analysis and guidelines. J Med Ethics. 2016 Dec;42(12):776-783. doi: 10.1136/medethics-2015-103333. Epub 2016 Oct 24. PMID 27777269
- [Derived] Wartolowska K, Collins GS, Hopewell S, Judge A, Dean BJ, Rombach I, Beard DJ, Carr AJ. Feasibility of surgical randomised controlled trials with a placebo arm: a systematic review. BMJ Open. 2016 Mar 15;6(3):e010194. doi: 10.1136/bmjopen-2015-010194. PMID 27008687
- [Derived] Beard D, Rees J, Rombach I, Cooper C, Cook J, Merritt N, Gray A, Gwilym S, Judge A, Savulescu J, Moser J, Donovan J, Jepson M, Wilson C, Tracey I, Wartolowska K, Dean B, Carr A; CSAW Study Group. The CSAW Study (Can Shoulder Arthroscopy Work?) - a placebo-controlled surgical intervention trial assessing the clinical and cost effectiveness of arthroscopic subacromial decompression for shoulder pain: study protocol for a randomised controlled trial. Trials. 2015 May 9;16:210. doi: 10.1186/s13063-015-0725-y. PMID 25956385
- [Derived] Wartolowska K, Beard DJ, Carr AJ. Attitudes and beliefs about placebo surgery among orthopedic shoulder surgeons in the United Kingdom. PLoS One. 2014 Mar 14;9(3):e91699. doi: 10.1371/journal.pone.0091699. eCollection 2014. PMID 24632880
- See also: Webpage — https://www.ndorms.ox.ac.uk/research/clinical-trials/completed-trials/csaw